CLINICAL TRIAL: NCT07223580
Title: Evaluating The Role Of Corticosteroids In Post-Ureteroscopy Recovery For Urinary Calculi
Brief Title: A Study Of Corticosteroid On Postoperative Pain After Ureteroscopy For Urinary Calculi
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karen L. Stern, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-003416
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Ureteroscopy; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care plus Corticosteroid (Experimental): Participants will receive standard of care postoperative ureteroscopy medication, with the addition of prednisone 25 mg.
  Interventions: Drug: Corticosteroid
- Standard of Care (Placebo Comparator): Participants will receive standard of care postoperative ureteroscopy medication, with the addition of a placebo pill.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Corticosteroid — In addition to the standard of care postoperative ureteroscopy medication, participants will be given prednisone 25 mg orally, once a day for 5 days post-surgery.
  Other Names: Prednisone
  Arms: Standard of care plus Corticosteroid
Other: Placebo — In addition to the standard of care postoperative ureteroscopy medication, participants will be given a placebo pill orally, once a day for 5 days post-surgery.
  Arms: Standard of Care

SUMMARY:
The purpose of this research is to evaluate if corticosteroid (prednisone) after ureteroscopy and placement of the stent will help alleviate postoperative pain control in addition to other normal postoperative pain medications

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with kidney or ureteral stones confirmed on imaging (CT of the abdomen or pelvis) and who elect for definitive treatment via ureteroscopy with placement of ureteral stent.
* Age 18 years or older
* Patients of either gender
* Patients of all ethnic backgrounds
* Cable of giving informed consent
* Capable and willing to fulfill the requirements of the study.

Exclusion Criteria:

* History of chronic pain
* Chronic use of opioids or other pain medication (>12 weeks)
* Known allergies to corticosteroids.
* Known or suspected pregnancy
* Inability to give informed consent or unable to meet requirements of the study for any reason.
* Bilateral ureteroscopy
* Current Corticosteroid Use
* Diabetic patients who are insulin dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale Pain Score | Baseline, Day 1 (Post-operatively), Day 2, Day 3
  Pain values reported by participants will be assessed using the 100-mm Visual Analogue Scale (VAS). The VAS line will be 100 mm long with no intermediate delineations. Each end will be marked with "no pain" on the left, and "worst possible pain" on the right. Participants will identify their pain level by indicating a point on the line between each end. That point will be measured from the "No pain" end, and the number of millimeters will be reported as the pain score.

SECONDARY OUTCOMES:
Number of times non-opioid analgesics medication used | 3 days
  Total number of times participants used non-opioid analgesics medication
Cumulative usage of non-opioid analgesics medication | 3 days
  Total use of non-opioid analgesics medication of any kind, reported in mg
Change in Wisconsin Stone Quality of Life Questionnaire (WISQOL) score | Day 2 (Post-operatively), Day 3
  The Wisconsin Stone Quality of Life (WISQOL) questionnaire is a 29 item survey that assesses quality of life for participants with kidney stones and covers four domains: social impact, emotional impact, stone-related symptom impact, and vitality. Questions are answered on a 5-point Likert scale, (1 = Very true, 5 = Not at all true), with a total maximum score of 140. Higher scores indicate a better quality of life.
Change in Canadian Endourology Group Stent Symptom Score (CEGSSS) score | Day 1 (Post-operatively), Day 2, Day 3
  The Canadian Endourology Group Stent Symptom Score (CEGSSS) is a 11-item questionnaire that assesses ureteral stent symptoms through three domains: urination, pain, and quality of life. Scoring is based on participant responses to the individual questions, with higher scores indicating a greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Stern, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials